CLINICAL TRIAL: NCT00026273
Title: Multicenter Phase III Open Label Randomized Trial Comparing CPT-11 In Combination With A 5-FU/FA Infusional Regimen To The Same 5-FU/FA Infusional Regimen Alone As Adjuvant Treatment Of Stage III Colon Cancer
Brief Title: Fluorouracil and Leucovorin With or Without Irinotecan in Treating Patients Following Surgery for Stage III Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: XRP 4174B-307; CDR0000069014; PFIZER-A5961053; RP-64174-V-307; EORTC-40993; PETACC-3
Record Dates: First submitted 2001-11-09; First posted 2003-08-05 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage III rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them after surgery may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of fluorouracil and leucovorin with or without irinotecan in treating patients who have undergone surgery for stage III colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free survival at 3 years of patients with resected stage III colorectal cancer treated with adjuvant fluorouracil and leucovorin calcium with or without irinotecan.
* Compare the disease-free and overall survival at 5 years of patients treated with these regimens.
* Compare the safety profiles of these treatment regimens in these patients.
* Compare the quality-adjusted survival of patients treated with these regimens.
* Correlate the expression of putative prognostic markers (thymidylate synthase, telomerase, topoisomerase) with disease-free and overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

Arm I

* Patients receive irinotecan IV over 30-90 minutes, leucovorin calcium IV over 2 hours, and fluorouracil IV over 24 hours weekly for 6 weeks. Courses repeat every 7 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* As an alternative schedule, patients may receive irinotecan IV over 30-90 minutes and day 1 and leucovorin calcium IV over 2 hours and fluorouracil IV over 22 hours on days 1 and 2 every 2 weeks for 6 weeks. Treatment repeats every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Arm II

* Patients receive leucovorin calcium and fluorouracil as in arm I. Quality of life may be assessed at baseline; prior to courses 2, 3, and 4; and at 1, 3, and 6 months.

Patients are followed every 3 months for 3 years and then every 6 months for 2 years.

PROJECTED ACCRUAL: Approximately 1800 patients (900 per arm) will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or intraperitoneal rectum

  * Stage III
  * Completely resected within the past 3-8 weeks

    * No gross or microscopic evidence of residual disease after surgery
* No rectal cancer requiring total meso-rectal resection or pre- or postoperative radiotherapy
* No prior curatively resected synchronous metastasis of colorectal cancer

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 150,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No myocardial infarction with the past year
* No uncontrolled hypertension
* No high-risk uncontrolled arrhythmia
* No unstable angina pectoris

Other:

* HIV negative
* No chronic diarrhea
* No current chronic inflammation or subobstruction of bowel after surgery
* No active uncontrolled infection
* No other prior or concurrent malignancy except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No psychological, social, familial, or geographical condition that would preclude follow-up
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior antineoplastic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics
* No prior celioscopic resection of primary tumor

Other:

* At least 30 days since prior participation in another clinical trial with any investigational drug
* No other concurrent experimental drugs
* No other concurrent anticancer therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01; Primary Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Cutsem, MD, PhD, Study Chair — University Hospital, Gasthuisberg
Locations (15):
- Allgemeines Krankenhaus der Stadt Wien, Vienna (Wien), Austria
- U.Z. Gasthuisberg, Leuven, Belgium
- National Cancer Institute of Egypt, Cairo, Egypt
- France (2):
  - CHU Pitie-Salpetriere, Paris
  - Hopital Tenon, Paris
- Universitats-Krankenhaus Eppendorf, Hamburg, Germany
- Italy (5):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Universita Degli Studi di Firenze - Policlin. di Careggi, Firenze (Florence)
  - Ospedale San Carlo Borromeo, Milano (Milan)
  - Azienda Ospedaliera S. Maria, Terni
  - Universita Degli Studi di Udine, Udine
- Instituto Portugues de Oncologia do Porto, Porto, Portugal
- Hospital Universarito "Reina Sofia", Córdoba, Spain
- Hopital Cantonal Universitaire de Geneva, Geneva, Switzerland
- Royal Marsden Hospital, Sutton, England, United Kingdom

REFERENCES:
- [Background] Punt CJ, Buyse M, Kohne CH, Hohenberger P, Labianca R, Schmoll HJ, Pahlman L, Sobrero A, Douillard JY. Endpoints in adjuvant treatment trials: a systematic review of the literature in colon cancer and proposed definitions for future trials. J Natl Cancer Inst. 2007 Jul 4;99(13):998-1003. doi: 10.1093/jnci/djm024. Epub 2007 Jun 27. PMID 17596575
- [Result] Roth AD, Tejpar S, Delorenzi M, Yan P, Fiocca R, Klingbiel D, Dietrich D, Biesmans B, Bodoky G, Barone C, Aranda E, Nordlinger B, Cisar L, Labianca R, Cunningham D, Van Cutsem E, Bosman F. Prognostic role of KRAS and BRAF in stage II and III resected colon cancer: results of the translational study on the PETACC-3, EORTC 40993, SAKK 60-00 trial. J Clin Oncol. 2010 Jan 20;28(3):466-74. doi: 10.1200/JCO.2009.23.3452. Epub 2009 Dec 14. PMID 20008640
- [Result] Bosman FT, Yan P, Tejpar S, Fiocca R, Van Cutsem E, Kennedy RD, Dietrich D, Roth A. Tissue biomarker development in a multicentre trial context: a feasibility study on the PETACC3 stage II and III colon cancer adjuvant treatment trial. Clin Cancer Res. 2009 Sep 1;15(17):5528-33. doi: 10.1158/1078-0432.CCR-09-0741. Epub 2009 Aug 18. PMID 19690194
- [Result] Roth AD, Tejpar S, Yan P, et al.: Correlation of molecular markers in colon cancer with stage-specific prognosis: results of the translational study on the PETACC 3 - EORTC 40993-SAKK 60-00 trial. [Abstract] American Society of Clinical Oncology 2009 Gastrointestinal Cancers Symposium, 15-17 January 2009, San Francisco, CA. A-288, 2009.
- [Result] Tejpar S, Bosman F, Delorenzi M, et al.: Microsatellite instability (MSI) in stage II and III colon cancer treated with 5FU-LV or 5FU-LV and irinotecan (PETACC 3-EORTC 40993-SAKK 60/00 trial). [Abstract] J Clin Oncol 27 (Suppl 15): A-4001, 2009.
- [Result] Van Cutsem E, Labianca R, Bodoky G, Barone C, Aranda E, Nordlinger B, Topham C, Tabernero J, Andre T, Sobrero AF, Mini E, Greil R, Di Costanzo F, Collette L, Cisar L, Zhang X, Khayat D, Bokemeyer C, Roth AD, Cunningham D. Randomized phase III trial comparing biweekly infusional fluorouracil/leucovorin alone or with irinotecan in the adjuvant treatment of stage III colon cancer: PETACC-3. J Clin Oncol. 2009 Jul 1;27(19):3117-25. doi: 10.1200/JCO.2008.21.6663. Epub 2009 May 18. PMID 19451425
- [Result] Roth AD, Yan P, Dietrich D, et al.: Does UGT1A1*28 homozygosity predict for severe toxicity in patients treated with 5-fluorouracil (5-FU)-irinotecan (IRI)? Results of the PETACC 3-EORTC 40993-SAKK 60/00 trial comparing IRI/5-FU/folinic acid (FA) to 5-FU/FA in stage II-III colon cancer. [Abstract] American Society of Clinical Oncology 2008 Gastrointestinal Cancers Symposium, 25-27 January 2008, Orlando, FL. A-277, 2008.
- [Result] Roth AD, Yan P, Dietrich D, et al.: Is UGT1A1*28 homozygosity the strongest predictor for severe hematotoxicity in patients treated with 5-fluorouracil (5-FU)-irinotecan (IRI)? Results of the PETACC 3 - EORTC 40993 -SAKK 60/00 trial comparing IRI/5-FU/folinic acid (FA) to 5-FU/FA in stage II- III colon cancer (COC) patients. [Abstract] J Clin Oncol 26 (Suppl 15): A-4036, 2008.
- [Result] van Cutsem E, Labianca R, Hossfeld D, et al.: Randomized phase III trial comparing infused irinotecan / 5-fluorouracil (5-FU)/folinic acid (IF) versus 5-FU/FA (F) in stage III colon cancer patients (pts). (PETACC 3). [Abstract] J Clin Oncol 23 (Suppl 16): A-LBA8, 3s, 2005.
- [Derived] Taieb J, Shi Q, Pederson L, Alberts S, Wolmark N, Van Cutsem E, de Gramont A, Kerr R, Grothey A, Lonardi S, Yoshino T, Yothers G, Sinicrope FA, Zaanan A, Andre T. Prognosis of microsatellite instability and/or mismatch repair deficiency stage III colon cancer patients after disease recurrence following adjuvant treatment: results of an ACCENT pooled analysis of seven studies. Ann Oncol. 2019 Sep 1;30(9):1466-1471. doi: 10.1093/annonc/mdz208. PMID 31268130
- [Derived] Klingbiel D, Saridaki Z, Roth AD, Bosman FT, Delorenzi M, Tejpar S. Prognosis of stage II and III colon cancer treated with adjuvant 5-fluorouracil or FOLFIRI in relation to microsatellite status: results of the PETACC-3 trial. Ann Oncol. 2015 Jan;26(1):126-132. doi: 10.1093/annonc/mdu499. Epub 2014 Oct 30. PMID 25361982